CLINICAL TRIAL: NCT05163730
Title: Clinical Evaluation of the Panbio™ COVID-19/ Flu A&B Rapid Panel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Rapid Diagnostics Jena GmbH (Industry)
Responsible Party: Sponsor
Organization: Abbott Rapid Dx (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SDRD-G-026-P
Record Dates: First submitted 2021-11-06; First posted 2021-12-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: COVID-19; Influenza A; Influenza Type B
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Panbio™ COVID-19/ Flu A&B Rapid Panel (Other): One nasal swab sample will be collected from both nostrils by operators and will be used to perform the Panbio™ COVID-19/ Flu A&B Rapid Panel test either in a laboratory or in a non-laboratory setting (e.g. GP centre or hospital clinic). Each Panbio™ COVID-19/ Flu A&B Rapid Panel result will be photographed by the observer at the time of test interpretation.
  Nasopharyngeal samples will be collected and used for RT-PCR testing as per local procedures.
  Nasal samples must always be collected prior to the Nasopharyngeal sampling.
  Interventions: Device: COVID-19/ Flu A&B Rapid Panel

INTERVENTIONS:
Device: COVID-19/ Flu A&B Rapid Panel — Rapid Diagnostic Device

SUMMARY:
This study is designed as a prospective, multicentric, clinical study to investigate the performance of the Panbio™ COVID-19/ Flu A&B Rapid Panel for the qualitative detection of COVID-19 antigen, Influenza A antigen (H1N1 and H3N2), and Influenza B antigen in human nasal swabs.

This study is part of the performance evaluation to support the CE conformity assessment procedures.

DETAILED DESCRIPTION:
After obtaining written informed consent, a study-specific participant identification number (ID) will be assigned to the participant. Participant demographics and a brief medical history will be collected.

One nasal swab sample will be collected from both nostrils by operators and will be used to perform the Panbio™ COVID-19/ Flu A&B Rapid Panel test either in a laboratory or in a non-laboratory setting (e.g. GP (general practitioner) centre or hospital clinic). Each Panbio™ COVID-19/ Flu A&B Rapid Panel result will be photographed by the observer at the time of test interpretation.

Nasopharyngeal samples will be collected and used for RT-PCR (Reverse transcription polymerase chain reaction) testing as per local procedures.

Nasal samples must always be collected prior to the Nasopharyngeal sampling. A minimum of 90 Flu A positive subjects, a minimum of 90 Flu B positive subjects and a minimum of 100 SARS-CoV-2 positive subjects will be enrolled. In addition, a minimum of 385 negative subjects will be enrolled.

In total, a minimum of 665 male and female subjects will be prospectively enrolled at multiple clinical sites.

Collection procedure will be a mid-turbinate nasal swab (deep nasal swab), by turning the swab five times in each nostril. Nasal samples must be collected prior to the Nasopharyngeal sampling.

The collected swab will be tested with the Panbio™ COVID-19/ Flu A&B Rapid Panel at the study site. Tubes and swabs should be labelled with the patient ID.

After the nasal sampling, study staff personnel will also collect one nasopharyngeal swab. The nasopharyngeal swab will be eluted in Universal Transport Media (UTM) and used for testing with RT-PCR protocols for Flu A, Flu B and SARS-CoV-2 as per local procedures.

The RT-PCR methods used must have CE marking or FDA approval, with COVID-19 and Flu assay clearance for nasopharyngeal specimens. Nasopharyngeal sampling should be performed by trained healthcare professionals who routinely conduct nasopharyngeal sampling as part of their other standard of care and clinical duties.

Each operator who performs a Panbio™ COVID-19/ Flu A&B Rapid Panel test will fill out a user evaluation questionnaire once, to assess the usability of the device.

All other aspects of the Subject's care will remain the same with no deviation from prescribed practice.

ELIGIBILITY:
Inclusion Criteria:

* • Subjects from all age groups, able and willing to provide written informed consent or assent, suspected of having a respiratory viral infection consistent with COVID-19 and or Flu by their healthcare provider within the first seven days of the onset of symptoms, and presenting at least two of the following symptoms: fever, headache, extreme tiredness, dry cough, sore throat, runny or stuffy nose, muscle aches, loss of smell, loss of taste or shortness of breath, will be prospectively enrolled.

Exclusion Criteria:

* • Subject has had a nasal or a nasopharyngeal swab taken within the last 4 hours.

  * Subject has active nose bleeds or acute facial injuries/trauma
  * Subject has received a nasal vaccine (i.e., FluMist®) within the previous five (5) days.
  * Subject is currently taking or has taken an antiviral medication-i.e., Amantadine, Rimantadine, Relenza® (Zanamivir), Tamiflu® (Oseltamivir Phosphate), and Flumadine®-for influenza within the previous thirty (30) days.
  * Subject is currently enrolled in a study to evaluate an investigational drug.
  * Subject is unwilling or unable to provide informed consent.
  * Vulnerable populations as deemed inappropriate for study by the site's PI and/or reviewing REC (Research Ethics Committee).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2472 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity | 8 months
  Sensitivity of 70% is the target at the lower bound of the 95% confidence interval for SARS-CoV-2 and 70% for each Flu. The target specificity is 95% at the lower bound of the 95% confidence interval for each test line.

SECONDARY OUTCOMES:
Usability | 8 months
  The secondary objective of this study is to assess the usability of the Panbio™ Rapid Panel, as collected by trained healthcare workers.

CONTACTS AND LOCATIONS:
Locations (1):
- Urgent Care, Easley, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No